CLINICAL TRIAL: NCT00161668
Title: Prospective Observational Study of Mylotarg (Gemtuzumab Ozogamicin) in Usual Care
Brief Title: Study Evaluating Mylotarg (Gemtuzumab Ozogamicin) in Usual Care
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0903X-100847
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Gemtuzumab

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Mylotarg

SUMMARY:
This study is designed to assess the safety of Mylotarg therapy in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Treated by Mylotarg
* Provide ICF

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (52):
- United States (52):
  - Tucson, Arizona
  - Berkely, California
  - Burbank, California
  - Concord, California
  - Loma Linda, California
  - Los Angeles, California
  - San Francisco, California
  - Sylmar, California
  - Denver, Colorado
  - Boynton Beach, Florida
  - Plantation, Florida
  - Stuart, Florida
  - Tamarac, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Shrevport, Louisiana
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Columbia, Missouri
  - St Louis, Missouri
  - Neptune City, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - The Bronx, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Temple, Texas
  - Arlington, Virginia
  - Richmond, Virginia
  - Charleston, West Virginia
  - Morgantown, West Virginia
  - Appleton, Wisconsin